CLINICAL TRIAL: NCT05909670
Title: FASTT Telehealth Behavioral Support Service for Caregivers of Children With Developmental Delay or Disability
Acronym: FASTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: Special X Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R41HD111097 (NIH)
Record Dates: First submitted 2023-05-12; First posted 2023-06-18 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Parent-Child Relations; Parenting; Child Behavior; Development Delay; Developmental Disability; Development Disorder, Child
Keywords: caregiving; family navigation; child-centered; strength-based; telehealth; text-based support
MeSH Terms: conditions — Child Behavior; Learning Disabilities; Developmental Disabilities

STUDY DESIGN:
Intervention Model Description: Caregivers of children will complete pre- and post-program assessments to determine the feasibility and acceptability of the intervention and exploratory effects on self-reported parenting stress and parenting sense of competence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase 1 intervention (Experimental): Families will receive text and telephone support for child behavior and parenting stress issues.
  Interventions: Behavioral: Family Advice and Support Text and Telephone (FASTT) program

INTERVENTIONS:
Behavioral: Family Advice and Support Text and Telephone (FASTT) program — The Family Advice Support Text and Telephone (FASTT) service is a telehealth model that provides on-demand, evidence-based advice and support to reduce child behavior problems, address concerns about child development, and help manage stress for caregivers of children with DD. By using text and telephone, which are widely available without disparities in access by race, ethnicity, or socioeconomic status, FASTT overcomes barriers associated with videoconferencing which requires dependable Internet and familiarity with technology use. FASTT allows support to be delivered at times and locations that are convenient for the caregiver.

SUMMARY:
Over 7 million children in the U.S. receive support for a developmental delay or disability (DD). For caregivers of these children, behavior issues that often accompany their child's condition create high levels of stress leading to increased mental and physical health issues and impacts on caregiver-child interactions and family functioning. Although evidence-based practices exist to help caregivers with their child's behavioral development, access to these services is often limited by rigid delivery models requiring in-person visits that can delay support and further increase the burden on families. These barriers are disproportionately higher for families of color and for those in low resource situations: an effect that has been exacerbated by reductions in services due to coronavirus disease 2019 (COVID-19). The overall objective of this project is to develop and implement a telehealth delivery model of rapid-response, evidence-based behavioral support to be provided in conjunction with an existing family navigation program (Undivided) serving parents of children with DD to create a commercially marketable product that will reduce barriers to services in local communities across the country.

This project will test the feasibility and acceptability of the Family Advice Text and Telephone (FASTT) support service for caregivers of young children. This Phase 1 application will enable a collaborative process to adapt evidence-based behavioral support to the specific needs of families of children ages birth to 12 with DD and integrate that support within the existing family navigation service. The rationale for the work is that providing effective, personalized support through the widely accessible mediums of text and telephone will get caregivers the help they need when and where they have time to access it and close in time to the behavioral issues they need help with, thus reducing caregiver stress and increasing their sense of competence and positive interactions with their child. Aim 1 determines the feasibility of delivering evidence-based behavioral support to caregivers of children with disabilities using on-demand text messaging. Aim 2 gauges the acceptability of the text-based support service to caregivers. Aim 3 assesses the extent to which text-based support reduces caregiver stress, improves caregiver sense of competence, and builds more positive perceptions of their child's behavior and their relationship with their child.

DETAILED DESCRIPTION:
The first three months of the project period will be used for planning and development, including cultural, content, and logistic adaptation and development of the evaluation procedures. During the next seven months, the adapted service will be implemented. The remaining two months of the project will be used for analysis of the evaluation data and creating the final report.

Implementation Plan. Integrating FASTT into the Undivided service platform will leverage the existing infrastructure and procedures of Undivided to link for families to FASTT Support Specialists. The Undivided infrastructure uses dedicated Care Navigators to assess family needs, provide assistance and encouragement in addressing those needs, and offer guidance and best practices to empower parents. The existing Undivided infrastructure uses a customized web-based and mobile app that provides messaging to the navigator support team for in-the-moment help and advice regarding service access and utilization, as well as a knowledgebase repository with expert-curated guides to support and navigation topics. Importantly, Undivided connects families to an online community of other caregivers of children with disabilities, effectively adding a peer support network for parents to share experiences, knowledge, and encouragement. The current Care Navigator team is focused on supporting families in accessing services, and stops short of making recommendations related to behavioral support.

Although family navigation services like Undivided have demonstrated efficacy in connecting families to services and reducing barriers to access, that function is dependent on the availability of services in the local community. Often, accessible services are not available to meet the needs of families due to insufficient capacity or the lack of flexible delivery methods. While availability of services has been an ongoing challenge for early intervention, it has been exacerbated by the advent of coronavirus disease 2019 (COVID-19) pandemic restrictions that reduced staffing and curtailed in-person support. These reductions have had significant negative effects on child behavior and caregiver stress and have disproportionately impacted families of color or those in low-resource circumstances. The FASTT service provides families with immediate expertise and support based on established principles of child development.

Undivided Care Navigators receiving support requests through the online app will identify family needs that fit within the FASTT scope of support. The FASTT scope focuses on three areas: 1) reducing child behavior problems, including sleep, feeding difficulties and picky eating, fearfulness, fussiness, tantrums, and defiant behavior; 2) addressing concerns about child development, including understanding what is typical vs. delayed development, having appropriate developmental expectations, knowing when to seek specialized support, and understanding how to promote healthy development through scaffolding; and 3) managing parenting stress, including maintaining work/life balance issues, regulating emotions, and reducing stress arising from concerns about attachment and parent/child relationship issues.

Caregivers requesting support in these areas will be provided with the FASTT line number which they can text to connect with a live Support Specialist. After a caregiver connects, they will be given the opportunity to continue the conversation by text or switch to a phone call at their preference. The Support Specialist begins with a set of discovery questions to understand the support topic, information about the strengths and challenges of the child, a history of the behavior, and what the caregiver has already tried to address the topic. Next, the Support Specialist suggests tips and advice drawn from established evidence-based practices (EBP) strategies and probes to determine the level of acceptance the caregiver has with the strategies. Motivational interviewing practices are used to support caregivers in selecting strategies that they feel they can implement. Recommendations are purposefully designed to be easily incorporated into caregivers' demanding schedules of tasks and activities. Conversations range from a few minutes to an hour or longer and can extend to days or weeks as caregivers may pause the conversation and return later when time is available. Strategies employ a strength-based approach that helps caregivers simultaneously facilitate skill development and diminish unwanted behaviors for their child. Parents can reach back out at any point for additional support or to share progress.

Experimental Design and Assessment Plan. This project will employ descriptive reporting of feasibility and acceptability, and quantitative analysis using a single-group pre and post program design. The primary outcomes of interest will be for feasibility and acceptability (see Table 1). Exploratory outcomes will include preliminary indications of impact on parenting stress and sense of competence, both general and for the specific topic of behavior support. Feasibility measures will include number of families who engaged in the service as a percent of those offered participation, the total number of sessions delivered, and characteristics of the sessions (e.g. length of text exchanges, span of case resolution in minutes or days, follow-up sessions on the same topic, and follow-up sessions on a different topic). Feasibility assessment will also include feedback from Undivided Care Navigators on ease of connecting families to the support and from the FASTT Support Specialists on ease and perceived efficacy of delivering support sessions. Acceptability measures will capture post-program perceptions of caregivers' satisfaction with the service (e.g. usefulness of the content, ease of access, and acceptability of telehealth delivery). Quantitative analysis will include pre and post evaluations collected at the program level (i.e. measures collected before and approximately two weeks after participating the in the FASTT program) and at the session level (i.e. brief measures collected at the beginning and end of support sessions). Pre-program assessment will include caregiver and family demographics (race/ethnicity, socioeconomic status, employment, developmental delay or disability of their child), general perceptions of parenting stress, parenting sense of competence, the topic of behavior or development they want support with (including frequency and intensity of challenging behaviors), and their stress and perceived self-efficacy around the specific behavior. Post-program assessment will include the same measures of general parenting stress and sense of competence, specific assessment of changes in stress and self-efficacy around the topic of the support session.

Data Analysis Plan. For Specific Aim 1, analysis will include descriptive numerical (e.g., mean, standard deviation, range) and visual depictions (e.g., histogram) of feasibility measures, including service engagement proportion, total number of delivered sessions, as well as session characteristics. We will also measure the metrics of support session delivery to enable future estimates of the cost of service provision.

For Specific Aim 2, we will first conduct descriptive numerical and visual depictions of acceptability measures of caregivers' satisfaction with the service (e.g., ratings of the degree to which participants found the program useful, easy to access, and respectful of their values). These acceptability measures are all based on a 1-to-7 rating scale, with "1" indicating extremely dissatisfied and "7" indicating extremely satisfied. To gauge the acceptability of this text-based support service, we will test the hypothesis that participants' average service satisfaction measures are all above 4 (indicating neither dissatisfied nor satisfied). Hypothesis testing will be performed using one-tail one-sample t-tests, although the non-parametric Wilcoxon signed-rank test will be used if the assumption of normality of the scores is not met. Sensitivity analyses in G*Power indicate that the proposed sample of 30 participants will allow us to detect a moderate-sized effect (Cohen's d = .46) with power of at least 0.80 (α = .05) in a one-tail one-sample t-test. With the one-tail non-parametric Wilcoxon signed-rank test, the proposed sample size of 30 will allow us to detect a moderate-sized effect (Cohen's d = .48) with power of .80 and α = .05.

For Specific Aim 3, exploratory analysis of impact measures will be performed using paired-sample t-tests to determine if post-program scores for parenting stress and parenting sense of competence significantly improve from corresponding pre-program scores (i.e., lower parenting stress, higher parenting sense of competence).If the assumption of normality of the scores is not met, the paired-sample non-parametric Wilcoxon signed-rank test will be used instead. Similar to hypothesis 2, sensitivity analyses in G*Power indicate that the proposed sample of 30 participants will allow us to detect moderate-sized effects (Cohen's d = .46 for regular paired-sample t-tests; Cohen's d = .48 for Wilcoxon signed-rank test) with statistical power of 0.8 and α of .05.

Table 1. Summary of Measures

Type Measure Baseline Endpoint Primary Feasibility x Acceptability x

Secondary Caregiver Stress x x Caregiver Self-efficacy x x

Exploratory analysis will also be conducted to examine potential heterogeneity in outcome variables of feasibility, acceptability, and program impact outcomes that may be explained by family demographics or child DD type. Both of these analyses will only be used to assess the promise of an intervention effect. More rigorous tests of efficacy will be conducted in Phase 2. All assessments will be self-administered by families and staff via an online survey platform to provide ease of access and flexibility. An option will be available to have a research assistant administer the assessments for families for whom self-administered, Internet-based surveys may pose a barrier.

ELIGIBILITY:
Inclusion Criteria:

* Must be a caregiver of a child age birth to 12 years with a developmental delay or disability
* Must understand spoken and written English sufficiently to complete survey questions and engage in the support program
* Must live within the State of California (i.e. the service area for the family navigation service conducting the project).
* Must have access to a phone or other device with text or voice capability. Note: Internet access is not required.
* There is no age limit for inclusion in this study. Parents or caregivers who are themselves under the age of 18 are will be included if they meet the study eligibility, which includes being the caregiver of a child age birth to 12 years with a DD. In these instances, consent will be obtained from the caregiver's legal parent or guardian.

Exclusion Criteria:

* Exclusion will be based on failure to meet inclusion criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Service engagement percentage as assessed by recruitment and consent records | Through study completion: an average of 1 year.
  This measure will include the number of families who opted to engage in the program as a percentage of the total number of families offered participation.
Program acceptability rating questionnaire | Through study completion: an average of 1 year.
  This measure will be the average of 3 questionnaire items that assess caregivers' satisfaction with the service (e.g., ratings of the degree to which participants found the program useful, easy to access, and respectful of their values). Participant responses will be captured using 7-point Likert scale, with "1" indicating extremely dissatisfied and "7" indicating extremely satisfied.

SECONDARY OUTCOMES:
Parenting Stress Index 4 - Short Form (PSI) | Through study completion: an average of 1 year.
  The PSI is a 36-item parent self-report measure of parenting stress rated on a 5-point Likert scale (strongly agree to strongly disagree) to yield a total stress score from three subscales (Difficult Child, Parent-Child Dysfunctional Interaction, and Parent Distress).
Parenting Sense of Competency Scale (PSOC) | Through study completion: an average of 1 year.
  The PSOC is a parent self-report measure with 18 items rated on a 4-point Likert scale (strongly agree to strongly disagree).

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Peake, PhD, Principal Investigator — University of Oregon
Locations (2):
- United States (2):
  - Special X Inc., dba Undivided, Los Angeles, California
  - University of Oregon, Eugene, Oregon

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data collected from the study will be eligible for sharing externally
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Eligible individual participant data will be made available 1-year after the study is complete
Access Criteria: Individual participant data access requests must be approved by the study's Principal Investigator. Requests should include information about who will be given access to the individual participant data and what the individual participant data will be used for. If approved, a Data Use Agreement (DUA) will need to be completed between the University of Oregon and the institution where the individual participant data will be sent.

REFERENCES:
- [Background] Grant R, Isakson EA. Regional variations in early intervention utilization for children with developmental delay. Matern Child Health J. 2013 Sep;17(7):1252-9. doi: 10.1007/s10995-012-1119-3. PMID 22918713
- [Background] Lindly OJ, Chavez AE, Zuckerman KE. Unmet Health Services Needs Among US Children with Developmental Disabilities: Associations with Family Impact and Child Functioning. J Dev Behav Pediatr. 2016 Nov/Dec;37(9):712-723. doi: 10.1097/DBP.0000000000000363. PMID 27801721
- [Background] Neece C, McIntyre LL, Fenning R. Examining the impact of COVID-19 in ethnically diverse families with young children with intellectual and developmental disabilities. J Intellect Disabil Res. 2020 Oct;64(10):739-749. doi: 10.1111/jir.12769. Epub 2020 Aug 18. PMID 32808424
- [Background] Jeste S, Hyde C, Distefano C, Halladay A, Ray S, Porath M, Wilson RB, Thurm A. Changes in access to educational and healthcare services for individuals with intellectual and developmental disabilities during COVID-19 restrictions. J Intellect Disabil Res. 2020 Nov;64(11):825-833. doi: 10.1111/jir.12776. Epub 2020 Sep 17. PMID 32939917
- [Background] Razai MS, Oakeshott P, Kankam H, Galea S, Stokes-Lampard H. Mitigating the psychological effects of social isolation during the covid-19 pandemic. BMJ. 2020 May 21;369:m1904. doi: 10.1136/bmj.m1904. No abstract available. PMID 32439691
- [Background] Spinelli M, Lionetti F, Setti A, Fasolo M. Parenting Stress During the COVID-19 Outbreak: Socioeconomic and Environmental Risk Factors and Implications for Children Emotion Regulation. Fam Process. 2021 Jun;60(2):639-653. doi: 10.1111/famp.12601. Epub 2020 Sep 28. PMID 32985703
- [Background] Morgenstern J, Kuerbis A, Houser J, Levak S, Amrhein P, Shao S, McKay JR. Dismantling motivational interviewing: Effects on initiation of behavior change among problem drinkers seeking treatment. Psychol Addict Behav. 2017 Nov;31(7):751-762. doi: 10.1037/adb0000317. Epub 2017 Sep 28. PMID 28956934
- [Background] Rollnick S, Butler CC, Kinnersley P, Gregory J, Mash B. Motivational interviewing. BMJ. 2010 Apr 27;340:c1900. doi: 10.1136/bmj.c1900. No abstract available. PMID 20423957
- [Background] Dunst CJ, Raab M, Hamby DW. Contrasting approaches to the response-contingent learning of young children with significant delays and their social-emotional consequences. Res Dev Disabil. 2017 Apr;63:67-73. doi: 10.1016/j.ridd.2017.02.009. Epub 2017 Mar 6. PMID 28268201
- [Background] Mottron L. Should we change targets and methods of early intervention in autism, in favor of a strengths-based education? Eur Child Adolesc Psychiatry. 2017 Jul;26(7):815-825. doi: 10.1007/s00787-017-0955-5. Epub 2017 Feb 8. PMID 28181042
- [Background] Waters L, Sun J. Can a Brief Strength-Based Parenting Intervention Boost Self-Efficacy and Positive Emotions in Parents. International Journal of Applied Positive Psychology 2016; 1, 41-56. https://doi.org/10.1007/s41042-017-0007-x
- [Background] Haskett ME, Ahern LS, Ward CS, Allaire JC. Factor structure and validity of the parenting stress index-short form. J Clin Child Adolesc Psychol. 2006 Jun;35(2):302-12. doi: 10.1207/s15374424jccp3502_14. PMID 16597226
- [Background] Reitman D, Currier RO, Stickle TR. A critical evaluation of the Parenting Stress Index-Short Form (PSI-SF) in a head start population. J Clin Child Adolesc Psychol. 2002 Sep;31(3):384-92. doi: 10.1207/S15374424JCCP3103_10. PMID 12149976
- [Background] Zaidman-Zait A, Mirenda P, Zumbo BD, Wellington S, Dua V, Kalynchuk K. An item response theory analysis of the Parenting Stress Index-Short Form with parents of children with autism spectrum disorders. J Child Psychol Psychiatry. 2010 Nov;51(11):1269-77. doi: 10.1111/j.1469-7610.2010.02266.x. PMID 20546082
- [Background] Johnston C, Mash EJ. A measure of parenting satisfaction and efficacy. Journal of clinical child psychology 1989; 18, 167-175.
- [Background] Gerald B. A Brief Review of Independent, Dependent and One Sample t-test. International Journal of Applied Mathematics and Theoretical Physics 2018; 4, 50. https://doi.org/10.11648/j.ijamtp.20180402.13
- [Background] Lowry R. Subchapter 12a: The Wilcoxon signed rank test. VassarStats: Website for statistical computation. Retrieved July 2000; 20, http://facultysites.vassar.edu/lowry/PDF/c12a.pdf
- [Background] Marsden E, Torgerson CJ. Single group, pre- and post-test research designs: Some methodological concerns. Oxford Review of Education 2012; 38, 583-616. https://doi.org/10.1080/03054985.2012.731208